CLINICAL TRIAL: NCT02477007
Title: Phase III Clinical Trial Studying Analgesic Efficacy of Morphine Alone or Combined With Paracetamol and/or Ibuprofen for Long-bones Fractures in Children
Brief Title: Analgesic Efficacy of Morphine Alone or Combined With Paracetamol and/or Ibuprofen for Long-bones Fractures in Children
Acronym: MORPHAPAIN
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: URC-CIC Paris Descartes Necker Cochin (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Quadruple | Purpose: Treatment
Other Study IDs: P130921; 2015-001458-14 (EudraCT Number)
Record Dates: First submitted 2015-04-09; First posted 2015-06-22 (Estimated); Last update posted 2025-11-20 (Actual); Status verified 2025-10

CONDITIONS: Pain; Long-bone Fractures
Keywords: Paediatric emergency; pain; long-bones fractures; morphine; ibuprofen; paracetamol; children
MeSH Terms: conditions — Pain | interventions — Acetaminophen; Ibuprofen

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- Ibuprofen+placebo of paracetamol (Experimental): Patients will receive in addition to morphine (usual care) ibuprofen and placebo of paracetamol
  Interventions: Drug: Ibuprofen; Drug: Placebo
- Paracetamol + placebo of ibuprofen (Experimental): Patients will receive in addition to morphine (usual care) paracetamol and placebo of ibuprofen
  Interventions: Drug: Paracetamol; Drug: Placebo
- Paracetamol + ibuprofen (Experimental): Patients will receive in addition to morphine (usual care) paracetamol and ibuprofen
  Interventions: Drug: paracetamol + ibuprofen
- Placebo of paracetamol + placebo of ibuprofen (Placebo Comparator): Patients will receive morphine alone(usual care).
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Paracetamol — Paracetamol will be an oral solution of 30 mg/ml. The doses of paracetamol will be 15 mg/kg (maximum dose: 1g).
  Arms: Paracetamol + placebo of ibuprofen
Drug: Ibuprofen — Ibuprofen will be an oral suspension of 20mg/ml. The doses of ibuprofen 10 mg/kg (maximum dose: 400 mg).
  Arms: Ibuprofen+placebo of paracetamol
Drug: paracetamol + ibuprofen — Paracetamol will be an oral solution of 30 mg/ml. The doses of paracetamol will be 15 mg/kg (maximum dose: 1g) Ibuprofen will be an oral suspension of 20mg/ml. The doses of ibuprofen 10 mg/kg (maximum dose: 400 mg).
  Arms: Paracetamol + ibuprofen
Drug: Placebo — Placebo will have the closest flavour, smell and aspect to the active substances, respectively paracetamol and ibuprofen. Placebo will be prepared in bottles with a fake label of active substances for a better blinding both for the nurse and the patient. Labels will be hiding by a mask.
  Arms: Ibuprofen+placebo of paracetamol; Paracetamol + placebo of ibuprofen; Placebo of paracetamol + placebo of ibuprofen

SUMMARY:
The main objective of this study is to evaluate the efficacy of two drugs: paracetamol and ibuprofen in association with morphine, compared with morphine alone on analgesia in children seen in the emergency department for a long-bone fracture and also to study the potential synergic effect of the association paracetamol and ibuprofen.

DETAILED DESCRIPTION:
Long-bone fractures are a very common complain for visits in paediatric emergency departments. Since these fractures are often very painful, morphine is considered the cornerstone treatment in case of severe pain. Very few data are available concerning the assessment of analgesic treatment in this condition. In our previous study, less than 50% of patients with a limb fracture had a Visual Analog Scale (VAS) ≤ 30 mm after morphine administration. Thus, one study make the hypothesis that the use of a combination of morphine and/or paracetamol and/or NSAID could be an effective and safe option for the treatment of pain due to long bone fractures. We undertake to compare different combinations of paracetamol and ibuprofen with morphine to determine the efficacy and safety of these strategies in emergency department paediatric patients with acute traumatic limb pain.

The main objective of this study is to evaluate the efficacy of two drugs: paracetamol and ibuprofen in association with morphine, compared with morphine alone on analgesia in children seen in the emergency department for a long-bone fracture and also to study the potential synergic effect of the association paracetamol and ibuprofen.

Second objectives are

* to compare the long term analgesic efficacy of 4 analgesic regimens a)ibuprofen/morphine, b)paracetamol/morphine, c)ibuprofen/paracetamol/morphine and d)morphine for long bone fracture management in the paediatric emergency department.
* To assess the tolerance of these 4 regimens.

The study is considered as a success if children 2-6 years (6 years included) have a pain score Evendol < 5 and children 7-17 years (17 years included) have a pain score assessed by Visual Analog Scale (VAS) ≤ 30 without additional analgesic treatment 30 minutes after drug administration.

ELIGIBILITY:
Inclusion Criteria:

* children aged 2 through 17 years (17 years included)
* suspected fracture of a long bone requiring morphine analgesia (VAS ≥ 60/100 or Evendol ≥ 7/15 at the arrival at emergency department)
* within the first 12 hours after the injury
* at least one signed parental informed consent
* affiliated to health insurance

Exclusion Criteria:

* analgesic treatment within the 6 hours before inclusion
* contraindication to one of the experimental drug: Paracetamol or Ibuprofen
* contraindication to Morphine
* cognitive impairment
* multiple injuries
* resuscitation manœuvres
* suspected femur fracture
* open fracture
* pregnant women in the third trimester

Ages: 2 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 304 (Actual)
Dates: Start 2015-12-03 (Actual); Primary Completion 2018-11-21 (Actual); Study Completion 2018-11-21 (Actual)

PRIMARY OUTCOMES:
Degree of pain measured by the EVENDOL score | 30 minutes
  To evaluate the degree of pain for children between 2 years and 6 years included : Evendol scale is a validated pain scale for use in the accident and emergency departments on children under 7 years old. Success: children 2-6 years (6 years included) with a pain score Evendol < 5 without additional analgesic treatment at 30 minutes after drug administration (DA)
Degree of pain measured by the Visual Analog Scale | 30 minutes
  To evaluate the degree of pain for children between 7 years and 17 years included. Patients will be asked to rate their pain severity on a validated 100 mm horizontal or vertical visual analog scale (VAS) marked "no pain" and "most severe pain" at the low and high ends respectively. A standardized explanation will be given to participating children. Success: children 7-17 years with pain score assessed by Visual Analog Scale (VAS) ≤ 30, without additional analgesic treatment at 30 minutes after drug administration (DA)

SECONDARY OUTCOMES:
Degree of pain measured by the EVENDOL score | after immobilisation
  To evaluate the degree of pain for children between 2 years and 6 years included : Evendol scale is a validated pain scale for use in the accident and emergency departments on children under 7 years old.
Degree of pain measured by the EVENDOL score | 15 minutes
  To evaluate the degree of pain for children between 2 years and 6 years included : Evendol scale is a validated pain scale for use in the accident and emergency departments on children under 7 years old.
Degree of pain measured by the EVENDOL score | 60 minutes
  To evaluate the degree of pain for children between 2 years and 6 years included : Evendol scale is a validated pain scale for use in the accident and emergency departments on children under 7 years old.
Degree of pain measured by the EVENDOL score | 90 minutes
  To evaluate the degree of pain for children between 2 years and 6 years included : Evendol scale is a validated pain scale for use in the accident and emergency departments on children under 7 years old.
Degree of pain measured by the EVENDOL score | 120 minutes
  To evaluate the degree of pain for children between 2 years and 6 years included : Evendol scale is a validated pain scale for use in the accident and emergency departments on children under 7 years old.
Degree of pain measured by the Visual Analog Scale | after immobilisation
  To evaluate the degree of pain for children between 7 years and 17 years included. Patients will be asked to rate their pain severity on a validated 100 mm horizontal or vertical visual analog scale (VAS) marked "no pain" and "most severe pain" at the low and high ends respectively. A standardized explanation will be given to participating children.
Degree of pain measured by the Visual Analog Scale | 15 minutes
  To evaluate the degree of pain for children between 7 years and 17 years included. Patients will be asked to rate their pain severity on a validated 100 mm horizontal or vertical visual analog scale (VAS) marked "no pain" and "most severe pain" at the low and high ends respectively. A standardized explanation will be given to participating children.
Degree of pain measured by the Visual Analog Scale | 60 minutes
  To evaluate the degree of pain for children between 7 years and 17 years included. Patients will be asked to rate their pain severity on a validated 100 mm horizontal or vertical visual analog scale (VAS) marked "no pain" and "most severe pain" at the low and high ends respectively. A standardized explanation will be given to participating children.
Degree of pain measured by the Visual Analog Scale | 90 minutes
  To evaluate the degree of pain for children between 7 years and 17 years included. Patients will be asked to rate their pain severity on a validated 100 mm horizontal or vertical visual analog scale (VAS) marked "no pain" and "most severe pain" at the low and high ends respectively. A standardized explanation will be given to participating children.
Degree of pain measured by the Visual Analog Scale | 120 minutes
  To evaluate the degree of pain for children between 7 years and 17 years included. Patients will be asked to rate their pain severity on a validated 100 mm horizontal or vertical visual analog scale (VAS) marked "no pain" and "most severe pain" at the low and high ends respectively. A standardized explanation will be given to participating children.
Tolerance of ibuprofen | 15 minutes
  occurrence of abdominal pain or diarrhea or nausea or vomiting or digestive bleeding or itching or rash.
Tolerance of ibuprofen | 30 minutes
  occurrence of abdominal pain or diarrhea or nausea or vomiting or digestive bleeding or itching or rash.
Tolerance of ibuprofen | 60 minutes
  occurrence of abdominal pain or diarrhea or nausea or vomiting or digestive bleeding or itching or rash.
Tolerance of ibuprofen | 90 minutes
  occurrence of abdominal pain or diarrhea or nausea or vomiting or digestive bleeding or itching or rash.
Tolerance of ibuprofen | 120 minutes
  occurrence of abdominal pain or diarrhea or nausea or vomiting or digestive bleeding or itching or rash.
Tolerance of paracetamol | 15 minutes
  Occurrence of rash or hives or itching or swelling
Tolerance of paracetamol | 30 minutes
  Occurrence of rash or hives or itching or swelling
Tolerance of paracetamol | 60 minutes
  Occurrence of rash or hives or itching or swelling
Tolerance of paracetamol | 90 minutes
  Occurrence of rash or hives or itching or swelling
Tolerance of paracetamol | 120 minutes
  Occurrence of rash or hives or itching or swelling
Tolerance of morphine | 15 minutes
  heart and respiratory rates,
Tolerance of morphine | 30 minutes
  heart and respiratory rates,
Tolerance of morphine | 60 minutes
  heart and respiratory rates,
Tolerance of morphine | 90 minutes
  heart and respiratory rates,
Tolerance of morphine | 120 minutes
  heart and respiratory rates,
Tolerance of morphine | 15 minutes
  oxygen saturation
Tolerance of morphine | 30 minutes
  oxygen saturation
Tolerance of morphine | 60 minutes
  oxygen saturation
Tolerance of morphine | 90 minutes
  oxygen saturation
Tolerance of morphine | 120 minutes
  oxygen saturation
Tolerance of morphine | 15 minutes
  occurrence of consciousness nausea and vomiting or pruritus or drowsiness or dizziness
Tolerance of morphine | 30 minutes
  occurrence of consciousness nausea and vomiting or pruritus or drowsiness or dizziness
Tolerance of morphine | 60 minutes
  occurrence of consciousness nausea and vomiting or pruritus or drowsiness or dizziness
Tolerance of morphine | 90 minutes
  occurrence of consciousness nausea and vomiting or pruritus or drowsiness or dizziness
Tolerance of morphine | 120 minutes
  occurrence of consciousness nausea and vomiting or pruritus or drowsiness or dizziness

CONTACTS AND LOCATIONS:
Overall Officials: Hélène Chappuy, MD PhD, Principal Investigator — Study Principal Investigator
Locations (1):
- Paediatric emergency Armand Trousseau hospital, Paris, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Clark E, Plint AC, Correll R, Gaboury I, Passi B. A randomized, controlled trial of acetaminophen, ibuprofen, and codeine for acute pain relief in children with musculoskeletal trauma. Pediatrics. 2007 Mar;119(3):460-7. doi: 10.1542/peds.2006-1347. PMID 17332198
- [Background] Koller DM, Myers AB, Lorenz D, Godambe SA. Effectiveness of oxycodone, ibuprofen, or the combination in the initial management of orthopedic injury-related pain in children. Pediatr Emerg Care. 2007 Sep;23(9):627-33. doi: 10.1097/PEC.0b013e31814a6a39. PMID 17876251
- [Background] Morton NS, O'Brien K. Analgesic efficacy of paracetamol and diclofenac in children receiving PCA morphine. Br J Anaesth. 1999 May;82(5):715-7. doi: 10.1093/bja/82.5.715. PMID 10536549